CLINICAL TRIAL: NCT00435279
Title: A 31-Week, Efficacy, Safety and Tolerability Study of Eszopiclone 3 mg Co-administered With Venlafaxine in Subjects With Major Depressive Disorder (MDD) and Co-existing Insomnia
Brief Title: A Study of Eszopiclone Co-administered With Venlafaxine in Subjects With Major Depressive Disorder and Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 190-062
Record Dates: First submitted 2007-02-12; First posted 2007-02-14 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Major Depressive Disorder; Insomnia
Keywords: Insomnia; Depression; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Sleep Initiation and Maintenance Disorders; Depression | interventions — Eszopiclone; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eszopiclone (Experimental)
  Interventions: Drug: Eszopiclone; Drug: Venlafaxine
- Placebo (Experimental)
  Interventions: Drug: Placebo; Drug: Venlafaxine

INTERVENTIONS:
Drug: Eszopiclone — Eszopiclone 3 mg
  Other Names: Lunesta
  Arms: Eszopiclone
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Venlafaxine — Venlafaxine 75 mcg Weeks 1, 2, 29, and 30 Venlafaxine 150 mcg Weeks 3 through 28
  Other Names: Effexor

SUMMARY:
To evaluate the antidepressant effect of adjunctive treatment with Eszopiclone in subjects receiving venlafaxine for the treatment of Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, parallel-group study. The study consists of two groups of subjects with Major Depressive Disorder randomized to treatment with either eszopiclone 3 mg or placebo nightly at bedtime for 31 weeks beginning the night of Visit 2. In addition, all subjects will receive open-label treatment with venlafaxine. Safety and efficacy will be evaluated using clinical observations as well as physician and subject administered ratings scales. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be male or female between the ages of 18 and 64, inclusive, at the time of signing consent.
* Subjects must have a primary diagnosis of Major Depressive Disorder (MDD) by DSM-IV criteria (296.XX) as determined by the Mini International Neuropsychiatric Interview (M.I.N.I.).
* MDD must be the condition that was chiefly responsible for motivating the subject to seek treatment.
* Subjects must have a 17-item Hamilton Depression Scale (HAM-D-17) total score of > 22 at the screening visit.

Exclusion Criteria:

* Subjects who have a HAM-D-17 total score < 18 at Visit 2 will be discontinued from the study.
* All subjects who do not meet DSM-IV criteria (307.42) for Insomnia related to a Major Depressive Disorder.
* Subjects with less than a total sleep time < 6.5 hours at least three times per week over the past month.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 678 (Actual)
Dates: Start 2007-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change from baseline in HAM-D-17 total score at Week 8. | Week 8

SECONDARY OUTCOMES:
The key secondary endpoint is the change from baseline in the mean subjective Total Sleep Time (TST) during Week 1. | Week 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, CNS, Study Chair — Sumitomo Pharma America, Inc.
Locations (52):
- Austria (2):
  - Salzburg
  - Vienna
- Croatia (2):
  - Split
  - Zagreb
- France (9):
  - Arcachon
  - Caen
  - Élancourt
  - Le Pecq
  - Rennes
  - Savigny-sur-Orge
  - Strasbourg
  - Toulouse
  - Verasailles
- Hungary (4):
  - Balassagyarmat
  - Budapest
  - Cegléd
  - Nyíregyháza
- Poland (7):
  - Bełchatów
  - Bydgoszcz
  - Krakow
  - Lodz
  - Lublin
  - Torun
  - Tuszyn
- Romania (3):
  - Bucharest
  - Lasi
  - Oradea
- Russia (5):
  - Arkhangelsk
  - Belchatow
  - Moscow
  - Saint Petersburg
  - Stavropol
- Serbia (4):
  - Belgrade
  - Kragujevac
  - Niš
  - Novi Sad
- Ukraine (7):
  - Donetsk, Pobeda District
  - Crimea
  - Dnipro
  - Kiev
  - Lviv
  - Odesa
  - Vinnitsa
- United Kingdom (9):
  - Avon, Bath
  - Glasgow, Scotland
  - Coventry
  - Fowey
  - Glasgow
  - Harrow
  - Haywards Heath
  - Plymouth
  - Warks